CLINICAL TRIAL: NCT03175887
Title: Dorsolateral Versus Medial Prefrontal TMS for Depression
Brief Title: Investigational TMS Treatment for Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI's discretion due to needing to modify study protocol.
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Holtzheimer, Director of Mood Disorder Services, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D17107
Record Dates: First submitted 2017-05-03; First posted 2017-06-05 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Depression; Treatment Resistant Depression
Keywords: depression; trd; treatment-resistant depression; TMS
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Arm (Experimental): Participants will receive TMS. They will be randomized to either the left dorsolateral prefrontal cortex or the medial prefrontal cortex.
  Interventions: Device: TMS
- Treatment Arm (Other): After the experimental arm, if a patient was randomized to the medial prefrontal cortex during the experimental arm and it did not work for them, they have the option of returning for a session of TMS to the FDA-approved dorsolateral prefrontal cortex.
  If they were assigned to the dorsolateral prefrontal cortex, they are not eligible to return for another set of treatment.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Transcranial magnetic stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain to improve symptoms of depression.

SUMMARY:
This study is aimed to help us learn about the effects of Transcranial Magnetic Stimulation at the forehead versus the left side of the head for treatment of Treatment Resistant Depression.

DETAILED DESCRIPTION:
While transcranial magnetic stimulation (TMS) to the left dorsolateral prefrontal cortex (DLPFC) is an FDA approved treatment for depression, a growing and converging database suggests the medial prefrontal cortex (MPFC) may be even more critical to the neurobiology of depression and antidepressant treatment response. This study will compare the efficacy of high frequency transcranial madntic stimulation on these two sections of the brain.

ELIGIBILITY:
Inclusion Criteria:

* 21-70 years old
* inadequate response to one current antidepressant medication
* currently depressed

Exclusion Criteria:

* psychiatric comorbidities

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms measured by the 17-item Hamilton Depression Rating Scale | Change from baseline Hamilton-17 score to follow-up visit at 1 week after final TMS intervention.
  Depressive symptoms will be measured by the 17-item Hamilton Depression Rating Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- White River Junction VA Medical Center, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No